CLINICAL TRIAL: NCT07110233
Title: Prospective Phase 2 Trial of Yttrium-90 Radiation Segmentectomy for Unresectable Hepatocellular Carcinoma
Brief Title: Yttrium-90 Radiation Segmentectomy for Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, R. Peter Lokken, MD, MPH, Associate Professor of Clinical Radiology, University of California, San Francisco
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RLOKKEN-A
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma; Unresectable Hepatocellular Carcinoma; Hepatocellular Cancer; Hepatocellular Carcinoma Non-resectable
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group 1. TheraSphere® Yttrium-90 microspheres (Experimental): Participants with a single tumor measuring 2-5 cm will receive one dose of TheraSphere® >250 Gy, and ideally > 400 Gy at the treating physician's discretion. Participants will be monitored for safety and complete quality of life questionnaires.
  Interventions: Device: TheraSphere® Yttrium-90 microspheres; Other: Health Related Quality of Life Questionnaires (HRQOL)
- Group 2. TheraSphere® Yttrium-90 microspheres (Experimental): Participants with 2-3 tumors ≤ 3 cm in diameter (T2 disease) will receive one dose of TheraSphere® >250 Gy, and ideally > 400 Gy at the treating physician's discretion. Participants will be monitored for safety and complete quality of life questionnaires.
  Interventions: Device: TheraSphere® Yttrium-90 microspheres; Other: Health Related Quality of Life Questionnaires (HRQOL)

INTERVENTIONS:
Device: TheraSphere® Yttrium-90 microspheres — Administered intra-arterially
  Other Names: TheraSphere®; Yttrium-90 microspheres; Microspheres Radionuclide
Other: Health Related Quality of Life Questionnaires (HRQOL) — Surveys administered
  Other Names: HRQOL Questionnaires

SUMMARY:
This is a prospective, single-blinded, single-arm, open-label Phase II trial of trans-arterial radiation segmentectomy using Yttrium-90 glass microspheres (TheraSphere®) for Hepatocellular Carcinoma (HCC) participants with unresectable Barcelona clinic liver cancer (BCLC) stage A disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the objective response rate (ORR) after radiation segmentectomy in participants with BCLC Stage A HCC and 1) a single solitary tumor measuring 2-5 centimeters (cm) and 2) 2 or 3 lesions each ≤ 3 cm.

II. To assess the safety of radiation segmentectomy.

SECONDARY OBJECTIVES:

I. To evaluate transplant-free survival.

II. To evaluate progression-free survival.

III. To evaluate the quality of life of participants.

IV. To evaluate the best imaging response. V. To determine the proportion of participants who remain active on the wait list for liver transplant and eventually are transplanted.

VI. The evaluate the number of participants that need additional treatment after TheraSphere® administration.

VII. Complete pathologic response (CPN) on liver explants among participants who underwent liver transplant.

Participants will undergo a single TheraSphere® administration and followed for quality-of-life outcomes and survival for up to 3 years after treatment. Participants will be censored at time of future transplant or if death occurs at any time after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically or imaging-confirmed confirmed HCC.
2. Group 1: Solitary tumor measuring 2-5 cm Or Group 2: 2-3 tumors each ≤ 3 cm in diameter.
3. No prior therapy to target tumor(s).
4. Not a candidate for surgical resection or thermal ablation after multidisciplinary assessment.
5. Age ≥22 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status = 0 or 1.
7. Demonstrated adequate organ function as defined below:

   1. Total bilirubin ≤3.0 mg/dL, unless elevated due to Gilbert's syndrome and direct bilirubin is within normal limits.
   2. aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) ≤5 X institutional upper limit of normal.
   3. alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) ≤5 X institutional upper limit of normal.
   4. Creatinine Glomerular filtration rate (GFR) > 30 ml/min.
8. Child-Pugh score ≤ B7
9. Albumin-bilirubin (ALBI) score 1-2
10. Participants who have received systemic therapy for HCC will be excluded from the trial.
11. Ability to understand a written informed consent document, and the willingness to sign it.
12. Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
13. Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria:

1. Macrovascular tumor invasion or infiltrative appearance of hepatocellular carcinoma.
2. History of severe allergy to iodinated contrast agents despite appropriate premedication.
3. Is currently receiving any other anti-cancer agents and any previous therapy with a device that uses Y90 as the radioisotope.
4. Symptomatic heart failure or severe valvular insufficiency.
5. Symptomatic pulmonary hypertension or lung disease.
6. Symptomatic ascites.
7. Severe uncontrolled coagulopathy International Normalized Ratio (INR) ≥ 3.0 or Platelet ≤ 20,000.
8. Main vein thrombosis (portal vein, both bland and tumor thrombus). Note: Less than lobar portal vein thrombosis is allowable only if the thrombus is bland.
9. Pregnant women are excluded from this study because TheraSphere emits radiation with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with TheraSphere, breastfeeding should be discontinued if the mother is treated with TheraSphere.
10. Lung-shunt fraction (LSF) resulting in anticipated lung dose of >30 Gray (Gy).
11. History of sphincterotomy, biliary-enteric anastomosis, or other biliary tract instrumentation. Note: Prior cholecystectomy with or without bile duct exploration is permitted.
12. Tumor perfused by extrahepatic collateral arteries.
13. Prior partial hepatectomy.
14. Psychiatric illness, other significant medical illness, or social situation which, in the investigator's opinion, would limit compliance or ability to comply with study requirements.
15. History of or current extrahepatic cancer.
16. Pulmonary insufficiency (defined by an arterial oxygen pressure (Pa,O2) of < 60 mmHg, or oxygen saturation (Sa,O2) of < 90%).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by mRECIST | Up to 6 months
  The objective response rate (ORR) after radiation segmentectomy in participants will be evaluated using a modified Response Evaluation Criteria in Solid Tumors (mRECIST) based on the best tumor response where Complete Response (CR) is defined as the disappearance of any intratumoral arterial enhancement in all target lesions, Partial Response (PR) is defined as a 30% decrease in the sum of diameters of viable (enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions, Stable Disease (SD) is defined as any cases that do not qualify for either partial response or progressive disease, and Progressive Disease (PD) is defined as an increase of at least 20% in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since treatment started.
Percentage of participants with treatment-related adverse events | Up to 6 months
  The percentage of participants with grade 3 or greater, treatment-related adverse events as classified by NCI Common Terminology Criteria for Adverse Events (CTCAE) will be reported.

SECONDARY OUTCOMES:
Median time from TheraSphere administration to transplant | Up to 3 years
  Transplant-free survival is defined as the time to transplant in months from TheraSphere administration until transplant or death by any cause using the Kaplan-Meier estimator and 90% confidence intervals.
Median time to disease progression | Up to 3 years
  Progression-free survival is defined as the time to tumor progression (in-field, distant intrahepatic, extrahepatic) based on mRECIST in months from TheraSphere administration until disease progression or death by any cause using the Kaplan-Meier estimator and 90% confidence intervals will be reported.
Changes in mean Functional Assessment of Cancer Therapy - Hepatobiliary (FACT-Hep) survey results over time | Up to 6 months
  The FACT-Hep is a 45-item self-report instrument developed to assess health-related quality of life (HRQoL) in persons diagnosed with hepatobiliary cancers and consists of the Functional Assessment of Cancer Therapy scale (FACT-G) which is a 27-item questionnaire designed to measure four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being and also includes a Hepatobiliary Cancer Subscale (HCS) which consists of an additional 18-items focusing on disease-specific symptoms such as back and stomach pain, gastrointestinal issues, anorexia, weight loss, and jaundice. Each item response score ranges from 0 (not at all) to 4 (very much) with a total score range from 0-180. The higher the score, the better the HRQoL. The change in mean scores over time will be reported.
Changes in mean EuroQol five-dimensional Questionnaire (EQ-5D) survey results over time | Up to 6 months
  EQ-5D is a standardized instrument for measuring generic health status. The health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The respondents self-rate their level of severity for each dimension by selecting one of the following responses: no problems (0), slight problems (1), mild problems (2), moderate problems (3), or severe problems (4) with a particular dimension. Lower scores indicate less issues/problems with that particular health dimension. The change in mean scores over time will be reported.
Best observed tumor response by mRECIST. | Up to 1 year
  Best imaging response at 1 year will be determined based on mRECIST criteria among imaging follow up within 1 year of treatment.
Proportion of participants on an active liver transplant waitlist who receive a transplant | Up to 3 years
  Participants status on the transplant list will be recorded and the proportion of them among all enrolled participants will be reported.
Proportion of participants requiring additional therapies | Up to 3 years
  The proportion of participants that need subsequent loco-regional therapies as deemed clinically indicated after TheraSphere administration will be reported.
Proportion of participants with Complete pathologic response (CPN) | Up to 3 years
  The proportion of participants who underwent a liver transplant and demonstrated CPN post-transplant will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Lokken, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No